CLINICAL TRIAL: NCT04138277
Title: A Phase 3 Open-label Extension Study to Assess the Long-term Safety and Efficacy of Intravenous ATB200 Co-administered With Oral AT2221 in Adult Subjects With Late-onset Pompe Disease (LOPD)
Brief Title: A Study to Assess the Long-term Safety and Efficacy of ATB200/AT2221 in Adult Subjects With Late-Onset Pompe Disease (LOPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATB200-07
Record Dates: First submitted 2019-10-18; First posted 2019-10-24 (Actual); Results first posted 2026-01-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pompe Disease (Late-onset)
Keywords: Pompe; rhGAA
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — miglustat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATB200/AT2221 (Experimental): Participants received ATB200 (cipaglucosidase alfa) co-administered with AT2221 capsule (miglustat)
  Interventions: Drug: AT2221; Biological: ATB200

INTERVENTIONS:
Drug: AT2221 — Participants received ATB200 co-administered with AT2221 (miglustat)
  Other Names: miglustat
Biological: ATB200 — Enzyme Replacement Therapy via intravenous infusion
  Other Names: cipaglucosidase alfa

SUMMARY:
This is a multicenter, international open-label extension study of ATB200/AT2221 in adult subjects with late-onset Pompe disease (LOPD) who completed Study ATB200-03.

DETAILED DESCRIPTION:
This is an open-label extension study for subjects who completed the ATB200-03 study. The subjects will stay in this study until regulatory approval or marketing authorization and/or commercialization in the participating subject's country.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have completed Study ATB200-03.

Note: Subjects who were forced to withdraw from Study ATB200-03 for a logistical reason not related to the efficacy or safety of cipaglucosidase alfa/miglustat (eg, hospitalization for a car accident, COVID-19 pandemic, or emergency surgery) that resulted in several consecutive missed doses may have been eligible to participate in this study upon approval by the Amicus medical monitor.

Exclusion Criteria

1. Subject plans to receive gene therapy or participate in another interventional study for Pompe disease.
2. Subject, if female, is pregnant or breastfeeding.
3. Subject, whether male or female, is planning to conceive a child during the study.
4. Subject had a hypersensitivity to any of the excipients in cipaglucosidase alfa or miglustat, or had a medical condition or any other extenuating circumstance that may have, in the opinion of the investigator or medical monitor, posed an undue safety risk to the subject or may have compromised his/her ability to comply with or adversely impacted protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (18):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - University of Florida Clinical Research Center, Gainesville, Florida
  - Emory Clinic, Atlanta, Georgia
  - IU Health Neuroscience Center, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Northwell Health, Great Neck, New York
  - NYU School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Gardner Neuroscience Institute, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Montefiore Clinical and Translational Research Center, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia
- Hospital Universitario Austral, Buenos Aires, Argentina
- Australia (4):
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
- Medizinische Universität Innsbruck, Innsbruck, Austria
- UZ Leuven, Leuven, Belgium
- University Clinical Centre of the Republic of Srpska, Banja Luka, The Republic of Srpska, Bosnia and Herzegovina
- Canada (2):
  - Alberta Children's Hospital, Heritage Medical Research Clinic, Calgary, Alberta
  - McMaster University Medical Centre, Hamilton, Ontario
- Aarhus Universitetshospital, Aarhus, Denmark
- France (5):
  - Hôpital Pierre Wertheimer, Bron
  - Hôpital Raymond Poincaré, Garches
  - Hôpital Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Pasteur 2, Nice
- Germany (3):
  - Universitätsklinikum Bonn, Bonn
  - Friedrich-Baur Institut, München
  - Universitätsklinikum Münster, Münster
- Eginition Hospital, Athens, Greece
- Hungary (3):
  - Semmelweis University, Budapest
  - University of Pécs, Pécs
  - University of Szeged, Szeged
- Italy (2):
  - UOC di Neurologia e Malattie Neuromuscolari, Messina
  - Universitaria Federico II, Napoli
- Japan (5):
  - Fukuoka University Hospital, Fukuoka
  - Kagoshima University Hospital, Kagashima
  - Izumi City General Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - The Jikei University Hospital, Tokyo
- Erasmus MC, Rotterdam, Netherlands
- University of Auckland, Auckland, New Zealand
- Centrum Medyczne Medyk, Rzeszów, Podkarpackie Voivodeship, Poland
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Pusan National University, Yangsan, Gyeongsangnam-do, South Korea
- Hospital de la Santa Creu I Sant Pau, Barcelona, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (4):
  - Queen Elizabeth Hospital Birmingham, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Free Hospital NHS Foundation Trust, London
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen H, Diaz-Manera J, Goker-Alpan O, Mozaffar T, Sitaraman Das S, Fox B, Amon F, O'Brien-Prince K, Goldman M, Holdbrook F, Jain V, Byrne BJ. Safety of home administration of cipaglucosidase alfa plus miglustat in late-onset Pompe disease: results from multiple clinical trials. Ther Adv Rare Dis. 2026 Jan 31;7:26330040261416943. doi: 10.1177/26330040261416943. eCollection 2026 Jan-Dec. PMID 41631150
- [Derived] Schoser B, Kishnani PS, Bratkovic D, Byrne BJ, Claeys KG, Diaz-Manera J, Laforet P, Roberts M, Toscano A, van der Ploeg AT, Castelli J, Goldman M, Holdbrook F, Sitaraman Das S, Wasfi Y, Mozaffar T; ATB200-07 Study Group. 104-week efficacy and safety of cipaglucosidase alfa plus miglustat in adults with late-onset Pompe disease: a phase III open-label extension study (ATB200-07). J Neurol. 2024 May;271(5):2810-2823. doi: 10.1007/s00415-024-12236-0. Epub 2024 Feb 28. PMID 38418563

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Continued Group: Participants who received ATB200 (20 mg/kg) co-administered with AT2221 (260 mg) in the feeder study who continued on that dose in this long-term extension
- Treatment Switched Group: Participants who received alglucosidase alfa/placebo in the feeder study who were switched to ATB200 (20 mg/kg) co-administered with AT2221 (260 mg) in this long-term extension
Period: Pretreatment
Arm/Group | Treatment Continued Group | Treatment Switched Group
Started | 82 | 37
Completed | 81 | 37
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Treatment
Arm/Group | Treatment Continued Group | Treatment Switched Group
Started | 81 | 37
Completed | 58 | 30
Not Completed | 23 | 7
Not completed — Adverse Event | 6 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Pregnancy | 3 | 0
Not completed — COVID-19 pandemic | 1 | 0
Not completed — Withdrawal by Subject | 9 | 3
Not completed — Sponsor decision | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Worsening of condition | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Continued Group | Treatment Switched Group | Total
Number analyzed (Participants) | 81 | 37 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 34 | 103
  >=65 years | 12 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (13.53) | 46.0 (13.47) | 48.0 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 18 | 66
  Male | 33 | 19 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 71 | 30 | 101
  More than one race | 5 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0
Enzyme Replacement Therapy (ERT)-experienced [Count of Participants; unit: Participants] | 61 | 29 | 90
ERT-naive [Count of Participants; unit: Participants] | 20 | 8 | 28
Age at diagnosis [Mean (Standard Deviation); unit: years] | 40.3 (13.82) | 37.2 (15.40) | 39.3 (14.35)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events (TEAEs), Treatment-emergent Serious Adverse Events (TESAEs), and TEAEs Leading to Discontinuation of Study Drug
Description: Number of subjects with TEAE, TESAE, and TEAE leading to discontinuation during this long-term extension study
Time Frame: Entire extension study (mean = 40.5 months on treatment)
Population: Open-label extension (OLE) Safety Population defined as all subjects who took at least one dose of ATB200/AT2221 combination treatment in Study ATB200-07
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 81 | 37
Participants
  Subjects with TEAEs | 80 | 37
  Subjects with TESAEs | 17 | 10
  Subjects with TEAEs leading to discontinuation | 6 | 2
  Subjects with TEAE leading to death | 1 | 0

2. Secondary Outcome: Change From Baseline in 6-Minute Walk Distance (6MWD)
Description: Motor function was measured using the 6-minute walk distance (meters)
Time Frame: baseline, Week 208
Population: Motor function was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 39 subjects in the Treatment Continued Group and 18 subjects in the Treatment Switched Group.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 39 | 18
meters | -33.3 (37.60) | -8.6 (62.77)

3. Secondary Outcome: Change From Baseline in Sitting % Predicted Forced Vital Capacity (FVC)
Description: Pulmonary function was measured by sitting % predicted forced vital capacity (FVC)
Time Frame: baseline, Week 208
Population: Pulmonary function was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 41 subjects in the Treatment Continued Group and 15 subjects in the Treatment Switched Group.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 41 | 15
percent predicted FVC | -3.8 (9.10) | -0.5 (8.54)

4. Secondary Outcome: Change From Baseline in Manual Muscle Testing (MMT) Lower Extremity Score
Description: Strength was measured by manual muscle testing (MMT) using the Medical Research Council grading scale (0 to 5 points, with 5 indicating normal function). Change from baseline values >0 represent improvement.
Time Frame: baseline, Week 208
Population: Muscle strength was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 35 subjects in the Treatment Continued Group and 15 subjects in the Treatment Switched Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 35 | 15
score on a scale | 0.6 (4.38) | 0.4 (2.61)

5. Secondary Outcome: Change From Baseline in the Total Score for Patient-reported Outcomes Measurement Information System (PROMIS®) - Physical Function
Description: Physical Function Short Form 20a (v2.0) consisted of 20 questions. The first 14 questions were each scored on a scale from 1 to 5 as follows: 1 = unable to do; 2 = with much difficulty; 3 = with some difficulty; 4 = with a little difficulty; 5 = without any difficulty; the next 6 questions were each scored on a scale from 1 to 5 as follows: 1 = cannot do; 2 = quite a lot; 3 = somewhat; 4 = very little; 5 = not at all. The total score was calculated by summing up scores (1 to 5) across all items. Total scores range from 20 to 100. A higher score represented a better outcome.
Time Frame: baseline, Week 208
Population: PROMIS-Physical Function was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 42 subjects in the Treatment Continued Group and 19 subjects in the Treatment Switched Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 42 | 19
score on a scale | -2.7 (8.38) | -2.5 (6.14)

6. Secondary Outcome: Change From Baseline in the Total Score for PROMIS® - Fatigue
Description: Fatigue Short Form 8a consisted of 6 questions, each scored on a scale from 1 to 5 as follows: 1 = not at all; 2 = a little bit; 3 = somewhat; 4 = quite a bit; 5 = very much; and 2 questions, each scored on a scale from 1 to 5 as follows: 1 = never; 2 = rarely; 3 = sometimes; 4 = often; 5 = always. The total score was calculated by summing up scores (1 to 5) across all items resulting in a total score range from 6 (minimum) to 30 (maximum). A lower score represented lower fatigue symptoms.
Time Frame: baseline, Week 208
Population: PROMIS-Fatigue was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 42 subjects in the Treatment Continued Group and 19 subjects in the Treatment Switched Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 42 | 19
score on a scale | 1.5 (7.14) | 1.1 (3.72)

7. Secondary Outcome: Change From Baseline in Gait, Stairs, Gower, Chair (GSGC) Test
Description: The GSGC consisted of a 10-meter walk for evaluation of gait, a 4-stair climb, Gowers' maneuver, and arising from a chair. Results of the GSGC included the time required to complete the individual tests, individual scores for each of the tests (1 to 7 points for each of gait, 4-stair climb, and Gowers' maneuver, and 1 to 6 points for arising from a chair), and a total score. GSGC total score was the sum of the component scores from the 4 functional tests. The total score ranged from a minimum of 4 points (normal performance) to a maximum of 27 points (worst performance).
Time Frame: baseline, Week 208
Population: GSGC was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 33 subjects in the Treatment Continued Group and 14 subjects in the Treatment Switched Group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 33 | 14
score on a scale | 0.5 (2.98) | 0.3 (1.59)

8. Secondary Outcome: Change From Baseline in EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) Responses
Description: The EuroQol 5 Dimensions 5 Levels (EQ-5D-5L) questionnaire comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: Level 1=no problems, Level 2=slight problems, Level 3=moderate problems, Level 4=severe problems, and Level 5=extreme problems. In this categorical assessment, subjects were asked to indicate their health state by ticking the box next to the most appropriate statement in each of the 5 dimensions.
  Outcomes for change from baseline at Week 208 include 'no change', 'worsening' relative to baseline category, or 'improvement' relative to baseline category. Changes (worsening or improvement) are shown by magnitude of change (how many Levels) in each categorical assessment.
Time Frame: baseline, Week 208
Population: EQ-5D-5L was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 42 subjects in the Treatment Continued Group and 19 subjects in the Treatment Switched Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 42 | 19
Participants
  Mobility: No change from baseline | 27 | 12
  Mobility: Worsening (1 level) | 4 | 1
  Mobility: Worsening (2 levels) | 0 | 0
  Mobility: Worsening (3 or 4 levels) | 0 | 0
  Mobility: Improvement (1 level) | 9 | 4
  Mobility: Improvement (2 levels) | 2 | 2
  Mobility: Improvement (3 or 4 levels) | 0 | 0
  Self-care: No change from baseline | 25 | 12
  Self-care: Worsening (1 level) | 5 | 4
  Self-care: Worsening (2 levels) | 0 | 0
  Self-care: Worsening (3 or 4 levels) | 0 | 0
  Self-care: Improvement (1 level) | 9 | 2
  Self-care: Improvement (2 levels) | 3 | 1
  Self-care: Improvement (3 or 4 levels) | 0 | 0
  Usual Activities: No change from baseline | 23 | 6
  Usual Activities: Worsening (1 level) | 5 | 6
  Usual Activities: Worsening (2 levels) | 1 | 0
  Usual Activities: Worsening (3 or 4 levels) | 0 | 0
  Usual Activities: Improvement (1 level) | 11 | 6
  Usual Activities: Improvement (2 levels) | 2 | 1
  Usual Activities: Improvement (3 or 4 levels) | 0 | 0
  Pain/discomfort: No change from baseline | 22 | 14
  Pain/discomfort: Worsening (1 level) | 8 | 1
  Pain/discomfort: Worsening (2 levels) | 0 | 2
  Pain/discomfort: Worsening (3 or 4 levels) | 0 | 0
  Pain/discomfort: Improvement (1 level) | 10 | 2
  Pain/discomfort: Improvement (2 levels) | 2 | 0
  Pain/discomfort: Improvement (3 or 4 levels) | 0 | 0
  Anxiety/depression: No change from baseline | 29 | 13
  Anxiety/depression: Worsening (1 level) | 4 | 1
  Anxiety/depression: Worsening (2 levels) | 1 | 0
  Anxiety/depression: Worsening (3 or 4 levels) | 0 | 0
  Anxiety/depression: Improvement (1 level) | 7 | 5
  Anxiety/depression: Improvement (2 levels) | 1 | 0
  Anxiety/depression: Improvement (3 or 4 levels) | 0 | 0

9. Secondary Outcome: Change From Baseline in Overall Physical Well-being (Subject's Global Impression of Change [SGIC], Question 1)
Description: The Subject's Global Impression of Change overall physical well-being (question 1) is scored on a 7-point rating scale ranging from "very much worse" to "very much improved."
Time Frame: baseline, Week 208
Population: The SGIC was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 42 subjects in the Treatment Continued Group and 19 subjects in the Treatment Switched Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 42 | 19
Participants
  Very much worse | 0 | 0
  Much worse | 0 | 1
  Somewhat worse | 12 | 2
  No change | 15 | 9
  Somewhat improved | 9 | 3
  Much improved | 4 | 3
  Very much improved | 2 | 1

10. Secondary Outcome: Change From Baseline in Physician's Global Impression of Change (PGIC) Overall Status
Description: The Physician's Global Impression of Change (PGIC) is designed to record the physician's assessment of the subject's status, taking into account the subject's signs and symptoms and other neuromuscular symptoms, and signs relative to their status at the Baseline Visit. The PGIC is based on a single item that is scored on a 7-point rating scale ranging from 1 "very much worse" to 7 "very much improved."
Time Frame: baseline, Week 208
Population: The PGIC was evaluated using the Full Analysis Set (consisting of subjects in the study who had both a valid baseline and at least 1 post-baseline assessment for at least 1 of the main efficacy endpoints). Baseline and Month 208 assessment available for 40 subjects in the Treatment Continued Group and 19 subjects in the Treatment Switched Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 40 | 19
Participants
  Very much worse | 0 | 0
  Much worse | 0 | 1
  Somewhat worse | 9 | 3
  No change | 21 | 8
  Somewhat improved | 6 | 5
  Much improved | 3 | 1
  Very much improved | 1 | 1

11. Secondary Outcome: Percent Change From Baseline in Creatine Kinase (U/L)
Description: Percent change from baseline to Week 208 in the levels of biomarker creatine kinase (CK)
Time Frame: baseline, Week 208
Population: The Full Analysis Set was used in analyses of biomarkers. A total of 40 subjects in the Treatment Continued Group and 18 subjects in the Treatment Switched Group had CK values at Week 208.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 40 | 18
percent change from baseline | -17.8 (27.93) | -29.0 (37.11)

12. Secondary Outcome: Percent Change From Baseline in Urine Hex4 (mmol/Mol Creatinine)
Description: Percent change from baseline to Week 208 in the levels of biomarker urine Hex4.
Time Frame: baseline, Week 208
Population: The Full Analysis Set was used in analyses of biomarkers. A total of 39 subjects in the Treatment Continued Group and 17 subjects in the Treatment Switched Group had urine hex4 values at Week 208.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 39 | 17
percent change from baseline | -16.7 (43.70) | -62.4 (17.80)

13. Secondary Outcome: Proportion of Subjects With Positive Anti-drug Antibodies at Baseline and Week 208
Description: Immunogenicity was assessed by the number (%) of subjects with positive specific anti-cipaglucosidase antibodies at baseline and at Week 208
Time Frame: baseline, Week 208
Population: In the Treatment Continued group, 76 subjects had immunogenicity data at baseline, and 41 subjects had data at Week 208. In the Treatment Switched group, 36 subjects had immunogenicity data at baseline and 20 subjects had data at Week 208.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Continued Group | Treatment Switched Group
Number analyzed (Participants) | 76 | 36
Participants
  Baseline | 63 | 30
  Week 208: number analyzed (Participants) | 41 | 20
  Week 208 | 34 | 17

ADVERSE EVENTS:
Time Frame: Adverse event data collected over duration of the study. Duration of participation varied by patient (range: 1 to 58 months).
Arm/Group | Treatment Continued Group | Treatment Switched Group
All-Cause Mortality (participants affected / at risk) | 1/81 | 0/37
Serious Adverse Events (participants affected / at risk) | 17/81 | 10/37
Other Adverse Events (participants affected / at risk) | 80/81 | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Continued Group (N=81) | Treatment Switched Group (N=37)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Conjunctival hemorrhage (Eye disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dementia with Lewy bodies (Nervous system disorders) | 1 | 0
Hypoesthesia (Nervous system disorders) | 1 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Continued Group (N=81) | Treatment Switched Group (N=37)
Anemia (Blood and lymphatic system disorders) | 2 | 2
Ear pain (Ear and labyrinth disorders) | 6 | 0
Diarrhea (Gastrointestinal disorders) | 21 | 7
Nausea (Gastrointestinal disorders) | 15 | 5
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Toothache (Gastrointestinal disorders) | 7 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 6 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 2
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 2
Fatigue (General disorders) | 13 | 8
Pyrexia (General disorders) | 9 | 2
Edema peripheral (General disorders) | 5 | 2
Pain (General disorders) | 4 | 2
Gait disturbance (General disorders) | 1 | 2
Adverse drug reaction (General disorders) | 0 | 2
COVID-19 (Infections and infestations) | 43 | 21
Nasopharyngitis (Infections and infestations) | 19 | 5
Urinary tract infection (Infections and infestations) | 12 | 4
Upper respiratory tract infection (Infections and infestations) | 11 | 5
Sinusitis (Infections and infestations) | 9 | 3
Influenza (Infections and infestations) | 8 | 1
Gastroenteritis (Infections and infestations) | 6 | 2
Lower respiratory tract infection (Infections and infestations) | 4 | 2
Rhinitis (Infections and infestations) | 4 | 5
Bronchitis (Infections and infestations) | 2 | 2
Pyuria (Infections and infestations) | 2 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 39 | 18
Vaccination complication (Injury, poisoning and procedural complications) | 15 | 4
Contusion (Injury, poisoning and procedural complications) | 9 | 10
Ligament sprain (Injury, poisoning and procedural complications) | 7 | 3
Limb injury (Injury, poisoning and procedural complications) | 5 | 6
Muscle strain (Injury, poisoning and procedural complications) | 6 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 5 | 2
Skin laceration (Injury, poisoning and procedural complications) | 4 | 2
Procedural pain (Injury, poisoning and procedural complications) | 2 | 3
SARS-CoV-2 test positive (Investigations) | 3 | 2
Hemoglobin decreased (Investigations) | 0 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2
Headache (Nervous system disorders) | 28 | 14
Dizziness (Nervous system disorders) | 6 | 2
Paraesthesia (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 1 | 3
Depression (Psychiatric disorders) | 8 | 0
Insomnia (Psychiatric disorders) | 3 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 | 1
Rash (Skin and subcutaneous tissue disorders) | 9 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 5 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 7 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT04138277/Prot_000.pdf
  • Statistical Analysis Plan (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04138277/SAP_001.pdf